CLINICAL TRIAL: NCT04752137
Title: Evaluation of Intraoperative Tumor Margin Identification With Fluorescent Dye Imaging
Brief Title: Intraoperative Tumor Margin Identification With ICG Dye Imaging
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Santiago Lozano-Calderon, Assistant Professor of Orthopaedic Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P003481
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Benign Neoplasm; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ICG Dye and use of SPY-PHI Imaging (Other): ICG will be administered in the pre-operative unit via IV injection at the time that they present to the pre-operative unit, which is approximately 4 hours before surgery. ICG Angiography (SPY PHI) will be performed to detect any residual signal
  Interventions: Drug: Indocyanine green; Device: SPY-PHI

INTERVENTIONS:
Drug: Indocyanine green — The SPY PHI and its dye Indocyanine Green dye (ICG) is a non-invasive device that is connected to a light source tower that is already available in the hospital in the operating room under Gynecology and Obstetrics Equipment. This is a special light source lamp that allows to test for vascularity in the soft tissues intraoperatively. Previous research in animal models proved the concept that the increased vascularity in tumors can be used to use this device to improve intraoperative assessment of tumor margins during resection. Our study will help to establish a correlation between activity with the dye and histological findings. This information has the potential to help sarcoma patients by avoiding staged surgeries, decreasing hospitalization times, and decreasing the likelihood of local recurrence by improving margin quality.
Device: SPY-PHI — The SPY PHI and its dye Indocyanine Green dye (ICG) is a non-invasive device that is connected to a light source tower that is already available in the hospital in the operating room under Gynecology and Obstetrics Equipment. This is a special light source lamp that allows to test for vascularity in the soft tissues intraoperatively. Previous research in animal models proved the concept that the increased vascularity in tumors can be used to use this device to improve intraoperative assessment of tumor margins during resection. Our study will help to establish a correlation between activity with the dye and histological findings. This information has the potential to help sarcoma patients by avoiding staged surgeries, decreasing hospitalization times, and decreasing the likelihood of local recurrence by improving margin quality.

SUMMARY:
In this research study we want to learn more about the use of indocyanine green (ICG) during bone or soft tissue mass resections. Indocyanine green (ICG) is a type of dye that is used in medical diagnostics. We want to determine if ICG-guided tumor resection is more effective in obtaining negative margins. Lastly, we want to assess traditional oncologic outcomes of local recurrence, time to metastatic disease, and overall and disease specific survival.

DETAILED DESCRIPTION:
If you are present for a preoperative clinic visit the day before your surgery, ICG may be administered via injection. Otherwise, ICG will be administered in the preoperative unit via IV injection at the time of presentation approximately 4 hours before your surgery. You will be monitored during and after ICG dosing.

During surgery ICG fluorescence using a near-infrared imager will be performed at the time of and immediately following primary tumor resection. The imager will evaluate the primary tumor to ensure appropriate tumor fluorescence. Once the primary resection is complete and the surgeon believes that he/she has achieved negative or planned positive margins, fluorescence measurements of the tumor bed will be performed. If areas of positive signal remain, these areas will be resected if possible and sent to pathology for histologic evaluation. It will be recorded if the surgeon perceived negative margins but the device detected positive margins.

Tumor specimens and residual fluorescence positive samples will be evaluated using fresh frozen and permanent histology. Permanent samples will be evaluated for tumor and local fluorescence using confocal microscopy with an ICG cube. Positive fluorescence signal and its correspondence with neoplasm will be noted, a will tumor that does not fluoresce.

Tissue being removed is 1-2 mm from non-structurally important tissue that either has or does not have signal positivity for additional pathologic assessment. It should have no impact on patient outcome, does not represent intervention on sensitive areas (such as neurovascular structures), and can further be used as potential margin around the tumor.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older who present to Massachusetts General Hospital Department of Orthopaedic Surgery with a benign or malignant bone or soft tissue mass that is consented for surgery during the study period.

Exclusion Criteria:

* Pregnant or nursing patients
* Patients with previously known anaphylaxis to IV contrast or iodine (other allergies may be considered on a case-by-case basis)
* Patients in renal failure who are not cleared for ICG administration by their primary physician or oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
image-guided prediction of local recurrence | 2 Years
  The primary outcome of this work is image-guided prediction of local recurrence, defined as pathologically confirmed return of the resected tumor local to the prior excision bed within 2 years of the primary surgery.

SECONDARY OUTCOMES:
Distant recurrence (metastatic disease) | 2 Years
  If a participant develops metastatic disease after surgery with ICG and SPY-PHI.
physician-perceived vs. device measured negative margins | 14 days
  physician-perceived vs. device measured negative margins (compared using pathologic specimens), which will be measured against formal margin analysis performed by a pathologist during the routine standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Lozano-Calderon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasif N. Comparative effectiveness research for sarcoma. Cancer Treat Res. 2015;164:51-65. doi: 10.1007/978-3-319-12553-4_4. PMID 25677018
- [Background] Fourman MS, Mahjoub A, Mandell JB, Yu S, Tebbets JC, Crasto JA, Alexander PE, Weiss KR. Quantitative Primary Tumor Indocyanine Green Measurements Predict Osteosarcoma Metastatic Lung Burden in a Mouse Model. Clin Orthop Relat Res. 2018 Mar;476(3):479-487. doi: 10.1007/s11999.0000000000000003. PMID 29408832
- [Background] Harati K, Lehnhardt M. The changing paradigm of resection margins in sarcoma resection. Innov Surg Sci. 2017 Dec 6;2(4):165-170. doi: 10.1515/iss-2017-0043. eCollection 2017 Dec. PMID 31579750
- [Background] Rath B, Hardes J, Tingart M, Braunschweig T, Eschweiler J, Migliorini F. [Resection margins in soft tissue sarcomas]. Orthopade. 2019 Sep;48(9):768-775. doi: 10.1007/s00132-019-03795-6. German. PMID 31463543
- [Background] Goertz O, Pieper A, Lohe LV, Stricker I, Dadras M, Behr B, Lehnhardt M, Harati K. The Impact of Surgical Margins and Adjuvant Radiotherapy in Patients with Undifferentiated Pleomorphic Sarcomas of the Extremities: A Single-Institutional Analysis of 192 Patients. Cancers (Basel). 2020 Feb 5;12(2):362. doi: 10.3390/cancers12020362. PMID 32033261
- [Background] Harati K, Goertz O, Pieper A, Daigeler A, Joneidi-Jafari H, Niggemann H, Stricker I, Lehnhardt M. Soft Tissue Sarcomas of the Extremities: Surgical Margins Can Be Close as Long as the Resected Tumor Has No Ink on It. Oncologist. 2017 Nov;22(11):1400-1410. doi: 10.1634/theoncologist.2016-0498. Epub 2017 Jul 24. PMID 28739867
- [Background] Fourman MS, Gersch RP, Levites HA, Phillips BT, Bui DT. Is There a Right Way to Interpret SPY? Normalization of Indocyanine Green Angiography Readings in a Burn Model. Plast Reconstr Surg. 2015 Jul;136(1):128e-130e. doi: 10.1097/PRS.0000000000001380. No abstract available. PMID 25803152
- [Background] Crasto JA, Fourman MS, Morales-Restrepo A, Mahjoub A, Mandell JB, Ramnath K, Tebbets JC, Watters RJ, Weiss KR. Disulfiram reduces metastatic osteosarcoma tumor burden in an immunocompetent Balb/c or-thotopic mouse model. Oncotarget. 2018 Jul 10;9(53):30163-30172. doi: 10.18632/oncotarget.25733. eCollection 2018 Jul 10. PMID 30046395
- [Background] Mahjoub A, Morales-Restrepo A, Fourman MS, Mandell JB, Feiqi L, Hankins ML, Watters RJ, Weiss KR. Tumor Resection Guided by Intraoperative Indocyanine Green Dye Fluorescence Angiography Results in Negative Surgical Margins and Decreased Local Recurrence in an Orthotopic Mouse Model of Osteosarcoma. Ann Surg Oncol. 2019 Mar;26(3):894-898. doi: 10.1245/s10434-018-07114-9. Epub 2018 Dec 27. PMID 30588559
- [Background] Gilg MM, Sunitsch S, Leitner L, Bergovec M, Szkandera J, Leithner A, Liegl-Atzwanger B. Tumor-associated mortality and prognostic factors in myxofibrosarcoma - A retrospective review of 109 patients. Orthop Traumatol Surg Res. 2020 Oct;106(6):1059-1065. doi: 10.1016/j.otsr.2020.04.017. Epub 2020 Aug 7. PMID 32778437
- [Background] Newton AD, Predina JD, Corbett CJ, Frenzel-Sulyok LG, Xia L, Petersson EJ, Tsourkas A, Nie S, Delikatny EJ, Singhal S. Optimization of Second Window Indocyanine Green for Intraoperative Near-Infrared Imaging of Thoracic Malignancy. J Am Coll Surg. 2019 Feb;228(2):188-197. doi: 10.1016/j.jamcollsurg.2018.11.003. Epub 2018 Nov 22. PMID 30471345
- [Background] Madajewski B, Judy BF, Mouchli A, Kapoor V, Holt D, Wang MD, Nie S, Singhal S. Intraoperative near-infrared imaging of surgical wounds after tumor resections can detect residual disease. Clin Cancer Res. 2012 Oct 15;18(20):5741-51. doi: 10.1158/1078-0432.CCR-12-1188. Epub 2012 Aug 29. PMID 22932668
- [Background] Holt D, Parthasarathy AB, Okusanya O, Keating J, Venegas O, Deshpande C, Karakousis G, Madajewski B, Durham A, Nie S, Yodh AG, Singhal S. Intraoperative near-infrared fluorescence imaging and spectroscopy identifies residual tumor cells in wounds. J Biomed Opt. 2015 Jul;20(7):76002. doi: 10.1117/1.JBO.20.7.076002. PMID 26160347